CLINICAL TRIAL: NCT05505604
Title: Comparison of Pericapsular Nerve Group Block (PENG) Versus Fascia Iliaca Compartment Block (FICB) for Hip Fracture Analgesia in Emergency Department Patients
Brief Title: PENG vs FICB for Hip Fracture in ED Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Matthew Kongkatong, MD, Assistant Professor of Emergency Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR220275
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Femoral Neck Fractures; Intertrochanteric Fractures
Keywords: PENG; FICB; Fascia Iliaca Compartment Block; Pericapsular Nerve Group Block; Hip fracture
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either a PENG or FICB. Baseline characteristics will be collected and NRS pain scores collected preblock and at specified time points post block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG (Active Comparator): Patients with hip fracture randomized to receive PENG block
  Interventions: Procedure: PENG
- FICB (Active Comparator): Patients with hip fracture randomized to received FICB
  Interventions: Procedure: FICB

INTERVENTIONS:
Procedure: PENG — patients will receive an ultrasound-guided Pericapsular Nerve Group Block with 20mL of 0.25% bupivacaine (not to exceed 2mg/kg)
  Arms: PENG
Procedure: FICB — Patients will receive an ultrasound-guided Fascia Iliaca Compartment Block with 20 mL of 0.25% bupivacaine (not to exceed 2 mg/kg) diluted to total volume of 40 mL of injectate
  Arms: FICB

SUMMARY:
Regional anesthesia for hip fractures has been shown to decrease rates of delirium in elderly patients with hip fractures as well as improve pain compared to systemic opioids. The Pericapsular Nerve Group (PENG) block has recently received attention as an alternative approach to femoral nerve block and Fascia Iliaca Compartment Block (FICB). The investigators seek to evaluate if there is a difference between the PENG and FICB in terms of efficacy of pain control in ED patients presenting with hip fracture. We hypothesize that the PENG block may be superior based on previous research.

DETAILED DESCRIPTION:
Fractures of the proximal femur are a common presentation to the emergency department and are an acutely painful condition. This condition predominantly affects elderly patients who are at risk for delirium and more susceptible to the adverse effects of systemic opioids. Regional anesthesia is an recommended component of pain control for elderly patients with hip fracture. The investigators seek to compare the efficacy of pain control of the Pericapsular Nerve Group (PENG) block with the Fascia Iliaca Compartment Block (FICB).

Previous studies have suggested that the PENG block may be superior to the FICB for pain control and results in less thigh motor weakness. The investigators will compare pain control (by difference in mean VAS score at set time points), systemic opioid use (in mean morphine equivalents prior to surgery), and motor function in patients with hip fractures who receive either block in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Proximal femur fracture

Exclusion Criteria:

* refusal to consent
* hemodynamic instability
* allergy to local anesthetics
* severe injury with instability
* severe medical conditions with instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 6 hours
  Median pain score on 0-10 Numeric Rating Scale

SECONDARY OUTCOMES:
Opioid use | From block administration until time of surgery or 24 hours if surgery performed >24 hours
  Mean opioid consumption in morphine equivalents

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Available from http://www.ncbi.nlm.nih.gov/books/NBK52651/ PMID 21413206
- [Background] Kim CH, Yang JY, Min CH, Shon HC, Kim JW, Lim EJ. The effect of regional nerve block on perioperative delirium in hip fracture surgery for the elderly: A systematic review and meta-analysis of randomized controlled trials. Orthop Traumatol Surg Res. 2022 Feb;108(1):103151. doi: 10.1016/j.otsr.2021.103151. Epub 2021 Nov 23. PMID 34826609
- [Background] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043
- [Background] Beaudoin FL, Haran JP, Liebmann O. A comparison of ultrasound-guided three-in-one femoral nerve block versus parenteral opioids alone for analgesia in emergency department patients with hip fractures: a randomized controlled trial. Acad Emerg Med. 2013 Jun;20(6):584-91. doi: 10.1111/acem.12154. PMID 23758305
- [Background] Fletcher AK, Rigby AS, Heyes FL. Three-in-one femoral nerve block as analgesia for fractured neck of femur in the emergency department: a randomized, controlled trial. Ann Emerg Med. 2003 Feb;41(2):227-33. doi: 10.1067/mem.2003.51. PMID 12548273
- [Background] Ketelaars R, Stollman JT, van Eeten E, Eikendal T, Bruhn J, van Geffen GJ. Emergency physician-performed ultrasound-guided nerve blocks in proximal femoral fractures provide safe and effective pain relief: a prospective observational study in The Netherlands. Int J Emerg Med. 2018 Mar 2;11(1):12. doi: 10.1186/s12245-018-0173-z. PMID 29500558
- [Background] Godoy Monzon D, Vazquez J, Jauregui JR, Iserson KV. Pain treatment in post-traumatic hip fracture in the elderly: regional block vs. systemic non-steroidal analgesics. Int J Emerg Med. 2010 Nov 6;3(4):321-5. doi: 10.1007/s12245-010-0234-4. PMID 21373300
- [Background] Reavley P, Montgomery AA, Smith JE, Binks S, Edwards J, Elder G, Benger J. Randomised trial of the fascia iliaca block versus the '3-in-1' block for femoral neck fractures in the emergency department. Emerg Med J. 2015 Sep;32(9):685-9. doi: 10.1136/emermed-2013-203407. Epub 2014 Nov 27. PMID 25430915
- [Background] Hong HK, Ma Y. The efficacy of fascia iliaca compartment block for pain control after hip fracture: A meta-analysis. Medicine (Baltimore). 2019 Jul;98(28):e16157. doi: 10.1097/MD.0000000000016157. PMID 31305398
- [Background] Hadzic A. Blocks for Hip Analgesia. In: Lopez AM, Balocco AL, Vandepitte C, Hadzic A, eds. Hadzic's Peripheral Nerve Blocks and Anatomy for Ultrasound-Guided Regional Anesthesia. 3rd ed. New York: McGraw Hill; 2022.
- [Background] Birnbaum K, Prescher A, Hessler S, Heller KD. The sensory innervation of the hip joint--an anatomical study. Surg Radiol Anat. 1997;19(6):371-5. doi: 10.1007/BF01628504. PMID 9479711
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962
- [Background] Mosaffa F, Taheri M, Manafi Rasi A, Samadpour H, Memary E, Mirkheshti A. Comparison of pericapsular nerve group (PENG) block with fascia iliaca compartment block (FICB) for pain control in hip fractures: A double-blind prospective randomized controlled clinical trial. Orthop Traumatol Surg Res. 2022 Feb;108(1):103135. doi: 10.1016/j.otsr.2021.103135. Epub 2021 Oct 29. PMID 34715388
- [Background] Fahey A, Cripps E, Ng A, Sweeny A, Snelling PJ. Pericapsular nerve group block for hip fracture is feasible, safe and effective in the emergency department: A prospective observational comparative cohort study. Emerg Med Australas. 2022 Dec;34(6):884-891. doi: 10.1111/1742-6723.14013. Epub 2022 Jun 14. PMID 35701386
- [Background] Allard C, Pardo E, de la Jonquiere C, Wyniecki A, Soulier A, Faddoul A, Tsai ES, Bonnet F, Verdonk F. Comparison between femoral block and PENG block in femoral neck fractures: A cohort study. PLoS One. 2021 Jun 4;16(6):e0252716. doi: 10.1371/journal.pone.0252716. eCollection 2021. PMID 34086782
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Jadon A, Mohsin K, Sahoo RK, Chakraborty S, Sinha N, Bakshi A. Comparison of supra-inguinal fascia iliaca versus pericapsular nerve block for ease of positioning during spinal anaesthesia: A randomised double-blinded trial. Indian J Anaesth. 2021 Aug;65(8):572-578. doi: 10.4103/ija.ija_417_21. Epub 2021 Aug 25. PMID 34584279
- [Background] Luftig J, Dreyfuss A, Mantuani D, Howell K, White A, Nagdev A. A new frontier in pelvic fracture pain control in the ED: Successful use of the pericapsular nerve group (PENG) block. Am J Emerg Med. 2020 Dec;38(12):2761.e5-2761.e9. doi: 10.1016/j.ajem.2020.05.085. Epub 2020 May 28. PMID 32532621
- [Background] Rocha-Romero A, Arias-Mejia K, Salas-Ruiz A, Peng PWH. Pericapsular nerve group (PENG) block for hip fracture in the emergency department: a case series. Anaesth Rep. 2021 May 18;9(1):97-100. doi: 10.1002/anr3.12118. eCollection 2021 Jan-Jun. PMID 34027410
- [Background] Gullupinar B, Saglam C, Unluer EE, Ayvat P, Ozturk K, Gul M, Tandon S. Effectiveness of pericapsular nerve group block with ultrasonography in patients diagnosed with hip fracture in the emergency department. Ulus Travma Acil Cerrahi Derg. 2022 Jun;28(6):832-838. doi: 10.14744/tjtes.2022.67817. PMID 35652877
- [Background] Lin DY, Morrison C, Brown B, Saies AA, Pawar R, Vermeulen M, Anderson SR, Lee TS, Doornberg J, Kroon HM, Jaarsma RL. Pericapsular nerve group (PENG) block provides improved short-term analgesia compared with the femoral nerve block in hip fracture surgery: a single-center double-blinded randomized comparative trial. Reg Anesth Pain Med. 2021 May;46(5):398-403. doi: 10.1136/rapm-2020-102315. Epub 2021 Feb 26. PMID 33637625
- [Background] Desmet M, Balocco AL, Van Belleghem V. Fascia iliaca compartment blocks: Different techniques and review of the literature. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):57-66. doi: 10.1016/j.bpa.2019.03.004. Epub 2019 Apr 17. PMID 31272654